CLINICAL TRIAL: NCT04115748
Title: A Phase 3, Randomized, Double-blind, Placebo and Adalimumab-controlled Study to Evaluate the Efficacy and Safety of Filgotinib in Subjects With Active Psoriatic Arthritis Who Are Naive to Biologic DMARD Therapy
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in Participants With Active Psoriatic Arthritis Who Are Naive to Biologic DMARD Therapy
Acronym: PENGUIN 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-431-4566; 2019-001996-35 (EudraCT Number); JapicCTI-205202 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — GLPG0634; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Filgotinib 200 mg (Main Study) (Experimental): Participants will receive filgotinib 200 mg + placebo to match (PTM) filgotinib 100 mg + PTM adalimumab injection for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab
- Filgotinib 100 mg (Main Study) (Experimental): Participants will receive PTM filgotinib 200 mg + filgotinib 100 mg + PTM adalimumab for up to 16 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab
- Adalimumab (Main Study) (Active Comparator): Participants will receive PTM filgotinib 200 mg + PTM filgotinib 100 mg + adalimumab 40 mg injection for up to 16 weeks.
  Interventions: Drug: Adalimumab; Drug: Placebo to match filgotinib
- Placebo (Main Study) (Placebo Comparator): Participants will receive PTM filgotinib 200 mg + PTM filgotinib 100 mg + PTM adalimumab injection for up to 16 weeks.
  Interventions: Drug: Placebo to match filgotinib; Drug: Placebo to match adalimumab
- Filgotinib 200 mg (Long Term Extension [LTE]) (Experimental): Participants will receive filgotinib 200 mg + PTM filgotinib 100 mg for up to 34 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Filgotinib 100 mg (LTE) (Experimental): Participants will receive PTM filgotinib 200 mg + filgotinib 100 mg for up to 34 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablets administered orally once daily with or without food
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg (LTE); Filgotinib 100 mg (Main Study); Filgotinib 200 mg (Long Term Extension [LTE]); Filgotinib 200 mg (Main Study)
Drug: Adalimumab — Injection administered subcutaneously once every 2 weeks
  Arms: Adalimumab (Main Study)
Drug: Placebo to match filgotinib — Tablets administered orally once daily with or without food
Drug: Placebo to match adalimumab — Injection administered subcutaneously once every 2 weeks
  Arms: Filgotinib 100 mg (Main Study); Filgotinib 200 mg (Main Study); Placebo (Main Study)

SUMMARY:
The primary objective of this study is to evaluate the effect of filgotinib compared to placebo as assessed by the American College of Rheumatology 20% improvement (ACR20) response in participants with active psoriatic arthritis who are naive to biologic disease-modifying anti-rheumatic drug (DMARD) therapy. The study consists of two parts, the Main Study and the Long Term Extension (LTE).

ELIGIBILITY:
Key Inclusion Criteria:

* Meet Classification Criteria for Psoriatic Arthritis (CASPAR) and have a history consistent with psoriatic arthritis (PsA) ≥ 6 months at Screening
* Have active PsA defined as ≥ 3 swollen joints (from a 66 swollen joint count [SJC]) and ≥ 3 tender joints (from a 68 tender joint count [TJC]) at Screening and Day 1; these may or may not be the same joints at Screening and Day 1
* Must have a documented history or active signs of at least one of the following at Screening:

  * Plaque psoriasis
  * Nail changes attributed to psoriasis
* Have had inadequate response or intolerance to ≥1 conventional synthetic disease-modifying anti-rheumatic drug (csDMARD), apremilast and / or NSAID, administered over the course of ≥ 12 weeks for the treatment of PsA, as per local guidelines / standard of care

Key Exclusion Criteria:

* Prior PsA or psoriasis treatment with a biologic DMARD
* Prior exposure to a janus kinase (JAK) inhibitor > 2 doses
* Any active / recent infection
* Any chronic and / or uncontrolled medical condition that would put the individual at increased risk during study participation or circumstances which may make an individual unlikely or unable to complete or comply with study procedures and requirements, per investigator judgement
* Any moderately to severely active musculoskeletal or skin disorder other than PsA or plaque psoriasis that would interfere with assessment of study parameters, as per judgement of investigator

NOTE: Prior history of reactive arthritis or axial spondyloarthritis is permitted if there is documentation of change in diagnosis to PsA or additional diagnosis of PsA

* Any history of an inflammatory arthropathy with onset before age 16 years old
* Active autoimmune disease that would interfere with assessment of study parameters or increase risk to the individual by participating in the study (e.g. uveitis, inflammatory bowel disease, uncontrolled thyroiditis, systemic vasculitis, transverse myelitis), per judgement of investigator
* Pregnancy or nursing females
* Active drug or alcohol abuse, as per judgement of investigator

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (74):
- United States (24):
  - Medvin Clinical Research, Covina, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Omega Research Debary, LLC, DeBary, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Hmd Research Llc, Orlando, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - ForCare Clinical Research, Tampa, Florida
  - BayCare Medical Group, Inc., Tampa, Florida
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Physician Research Collaaboration, LLCs, Lincoln, Nebraska
  - Atlantic Coast Research, Toms River, New Jersey
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Clinical Research Source Inc, Perrysburg, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Inc, dba, Columbia Arthritis Center, PA, Columbia, South Carolina
  - ACME Research, LLC, Orangeburg, South Carolina
  - Arthritis & Osteoporosis Clinic of Brazos Valley (Drug Shipment Address), College Station, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - West Virginia Research Institute PLLC, South Charleston, West Virginia
- Australia (3):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment - Plovdiv AD, Department Of Rheumatology, Plovdiv
  - Multiprofile Hospital for Active Treatment "Lyulin" EAD, Department of Rheumatology, Sofia
  - Diagnostic consultative center 17 Sofia EOOD, Sofia
  - "Medical center Synexus Sofia" EOOD, Sofia
  - "Medical center SYNEXUS SOFIA" EOOD, branch Stara Zagora, Stara Zagora
- G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Canada
- CCR Ostrava, s.r.o., Ostrava, Czechia
- Hungary (2):
  - Synexus (DRS) - Synexus Magyarorszag Kft. Budapest, Budapest
  - Synexus (DRS) - Synexus Magyarorszag Kft. Gyula, Gyula
- Japan (4):
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Daido Clinic, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Keio University Hospital, Tokyo
- New Zealand (4):
  - Waikato Hospital, Hamilton, WKO
  - Optimal Clinical Trials, Auckland
  - Capital & Coast District Health Board, Newtown
  - Clinical Trials Unit, Timaru Hospital, Timaru
- Poland (13):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok, Podlaskie
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela, Bydgoszcz
  - NSZOZ Unica CR, Dabrówka
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Malopolskie Badania Kliniczne SP Z O O Sp. k., Krakow
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Medycyna Kliniczna Marzena Waszczak-Jeka, Warsaw
  - Pheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Centrum Medyczne AMED Warszawa, Warsaw
  - REUMATOLOG WARSZAWA Specjalistyczna Praktyka Lekarska Dr n. med. Jakub Trefler, Warsaw
  - ARS RHEUMATICA Sp. Z.o.o., "REUMATIKA-Centrum Reumatologii", NZOZ, Warszawa, Mazowieckie
  - Centrum Medyczne Oporow, Wroclaw
- Russia (3):
  - Ulitsa Delegatskaya, 20, Building 1, Ulitsa Kasatkina, 7 Moscow, Russia, 127473/129301, Moskva
  - LLC "Biomed", Vladimir
  - Center for medical advice and research - PRACTICE LTD, Yaroslavl
- South Korea (3):
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Seoul National University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
- Spain (4):
  - Hospital Universitario 12 de Octubre, Avenida de Cordoba s/n, Rheumatology Service, Madrid, Spain, 28041, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Marques de Valdecilla, Rheumatology Service, Avda. Valdecilla s/n, Santander, Cantabria, 39008, Santander
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (7):
  - Buddhist Dalin Tzu Chi Hospital, Dailin Township
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Keelung Chang Gung Memorial Hospital, Keelung
  - Far Eastern Memorial Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Poland, the United States, Bulgaria, Spain, Australia, Japan, New Zealand, and Canada. The first participant was screened on 03 December 2019. The last study visit occurred on 11 May 2021.
Pre-assignment Details: 161 participants were screened.
Groups:
- Filgotinib 200 mg (Main Study): Filgotinib 200 milligrams (mg) tablet orally once daily + placebo to match (PTM) filgotinib 100 mg tablet orally once daily + PTM adalimumab subcutaneous (SC) injection every two weeks for 16 weeks.
- Filgotinib 100 mg (Main Study): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily + PTM Adalimumab SC injection every two weeks for 16 weeks.
- Adalimumab 40 mg (Main Study): PTM filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily + Adalimumab 40 mg SC injection every two weeks for 16 weeks.
- Placebo (Main Study): PTM filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily + PTM adalimumab SC injection every two weeks for 16 weeks.
- Filgotinib 200 mg From Filgotinib 200 mg (LTE): Long term extension (LTE):
  Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 34 weeks. Participants received filgotinib 200 mg in the Main Study.
- Filgotinib 100 mg From Filgotinib 100 mg (LTE): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for up to 34 weeks. Participants received filgotinib 100 mg in the Main Study.
- Filgotinib 200 mg From Adalimumab 40 mg (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 34 weeks. Participants received adalimumab 40 mg in the Main Study.
- Filgotinib 100 mg From Adalimumab 40 mg (LTE): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for up to 34 weeks. Participants received adalimumab 40 mg in the Main Study.
- Filgotinib 200 mg From Placebo (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 34 weeks. Participants received placebo in the Main Study.
- Filgotinib 100 mg From Placebo (LTE): Filgotinib 100 mg tablet orally once daily + PTM filgotinib 200 mg tablet orally once daily for up to 34 weeks. Participants received placebo in the Main Study.
Period: Main Study (Up to 16 Weeks)
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Adalimumab 40 mg (LTE) | Filgotinib 100 mg From Adalimumab 40 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Started | 19 | 19 | 9 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 16 | 7 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 15 | 16 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: LTE (After 16 Weeks to Week 50)
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Adalimumab 40 mg (LTE) | Filgotinib 100 mg From Adalimumab 40 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
Started | 0 (Participants who completed main study received filgotinib 200 mg.) | 0 (Participants who completed main study received filgotinib 100 mg.) | 0 (Participants who completed main study were randomized in LTE phase to receive filgotinib 200 mg or 100 mg.) | 0 (Participants who completed main study were randomized in LTE phase to receive filgotinib 200 mg or 100 mg.) | 4 (Participants who completed main study received filgotinib 200 mg.) | 3 (Participants who completed main study received filgotinib 100 mg.) | 1 (1 participant who received adalimumab injection and completed main study were randomised in LTE phase to receive filgotinib 200 mg.) | 1 (1 participant who received adalimumab injection and completed main study were randomised in LTE phase to receive filgotinib 100 mg.) | 2 (2 participants who received placebo and completed main study were randomised in LTE phase to receive filgotinib 200 mg.) | 2 (2 participants who received placebo and completed main study were randomised in LTE phase to receive filgotinib 100 mg.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 1 | 2 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib 200 mg (Main Study): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily + PTM adalimumab SC injection every two weeks for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study) | Total
Number analyzed (Participants) | 19 | 19 | 9 | 20 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13.4) | 46 (10.4) | 50 (10.4) | 47 (15.8) | 47 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 10 | 30
  Male | 10 | 12 | 5 | 10 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 18 | 19 | 9 | 19 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 18 | 18 | 8 | 20 | 64
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 9 | 9 | 5 | 11 | 34
  United States | 4 | 1 | 2 | 3 | 10
  Bulgaria | 3 | 3 | 0 | 1 | 7
  Spain | 1 | 2 | 1 | 3 | 7
  Australia | 1 | 2 | 0 | 1 | 4
  Japan | 0 | 1 | 1 | 0 | 2
  New Zealand | 1 | 1 | 0 | 0 | 2
  Canada | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement Response at Week 12
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: patient's global assessment of disease activity (PGADA) using a visual analogue scale (VAS) on a scale of 0 (very well) to 100 (very poor); physician's global assessment of disease activity (PHGADA) using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); health assessment questionnaire-disability index (HAQ-DI) inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain), and high-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all randomized participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adalimumab (Main Study): PTM filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily + Adalimumab 40 mg SC injection every two weeks for 16 weeks.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants | 76.8 [57.2 to 96.5] | 63.2 [38.8 to 87.5] | 67.2 [36.2 to 98.3] | 44.8 [22.8 to 66.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.048, Multiple imputation method — The stratification factors (Geographic Region, Concurrent Use of conventional synthetic (cs) DMARD(s) and/or Apremilast at Randomization, Prior Use of biologic (bio) DMARD(s)) and treatment groups were included in the imputation model as covariates; Difference in response rates = 32.1, 95% CI 2-sided [2.6 to 61.6]
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.23, Multiple imputation method — The stratification factors (geographic region, concurrent use of csDMARD(s) and/or apremilast at randomization, prior use of bioDMARD(s)) and treatment groups were included in the imputation model as covariates; Difference in response rates = 18.4, 95% CI 2-sided [-12.4 to 49.2]

2. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. It includes components of PGADA [using VAS on a scale of 0=very well to 100=very poor]; PhGADA [using VAS on a scale of 0=no disease activity to 100=maximum disease activity];36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains to determine a physical component summary (PCS) with a score range of 0-100, higher scores indicates better health status];TJC68;SJC66; leeds enthesitis index(LEI) [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis];Tender dactylitis count (TDC) [with a score range of 0 to 60, higher score indicates higher degree of dactylitis];C-reactive protein (CRP). Total score is calculated as the sum of the individual scores (each score adjusted by weighting factors). The score of PASDAS ranges from 0 to 10, lower scores indicates better function. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 5.9 (1.32) | 5.3 (0.99) | 5.5 (1.05) | 5.5 (1.05)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -1.5 (0.62) | -1.0 (0.99) | -1.3 (0.66) | -0.3 (0.80)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -2.5 (1.26) | -2.0 (1.48) | -2.6 (1.37) | -1.0 (1.04)

3. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) Response at Weeks 4, 8, 12, and 16
Description: MDA is a measure to indicate disease remission, and is based on a composite score of 7 domains. A participant is considered as having achieved the MDA if the participant fulfills at least 5 of the following 7 criteria: TJC68 ≤1; SJC66 ≤1; Psoriatic arthritis disease activity score (PASI) ≤1 for participants with psoriasis covering BSA <3% [PASI evaluates the severity and extent of psoriasis. In PASI, body is divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area is assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. The total score ranges from 0 (no disease) to 72 (maximal disease)]; patient's global assessment of PsA pain intensity (PGAPI) ≤15 [using VAS on a scale of 0 (no pain) to 100 (serious pain)]; PGADA ≤20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤0.5; LEI score ≤1 for participants with enthesitis at baseline.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 21.1 [0.1 to 42.0] | 16.7 [0.0 to 36.7] | 22.2 [0.0 to 54.9] | 5.0 [0.0 to 17.1]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 26.3 [3.9 to 48.7] | 31.6 [8.0 to 55.1] | 22.2 [0.0 to 54.9] | 15.8 [0.0 to 34.8]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 44.4 [18.7 to 70.2] | 47.4 [22.3 to 72.5] | 37.5 [0.0 to 77.3] | 15.8 [0.0 to 34.8]
  Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Week 16 | 27.8 [4.3 to 51.2] | 36.8 [12.5 to 61.2] | 37.5 [0.0 to 77.3] | 20.0 [0.0 to 40.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.17, Regression, Logistic — P-value was calculated by logistic regression with treatment group and stratification factors (geographic region and concurrent use of csDMARDs and/or apremilast at randomization) in the model; Difference in response rates = 16.1, 95% CI 2-sided [-9.7 to 41.9] — 95% confidence interval (CI) for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.27, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 11.7, 95% CI 2-sided [-13.3 to 36.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.42, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 10.5, 95% CI 2-sided [-20.4 to 41.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.26, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 15.8, 95% CI 2-sided [-16.0 to 47.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.062, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 28.7, 95% CI 2-sided [-5.0 to 62.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.047, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 31.6, 95% CI 2-sided [-1.5 to 64.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.58, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 7.8, 95% CI 2-sided [-24.6 to 40.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.27, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 16.8, 95% CI 2-sided [-16.2 to 49.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

4. Secondary Outcome: Percentage of Participants Who Achieved Very Low Disease Activity (VLDA) Response at Weeks 4, 8, 12, and 16
Description: VLDA is a measure to indicate disease remission, and is based on a composite score of 7 domains. A participant is considered as having achieved the VLDA if the participant fulfills all the seven criteria: TJC68 ≤1; SJC66 ≤1; PASI score ≤1 for participants with psoriasis covering BSA <3% [PASI evaluates the severity and extent of psoriasis. In PASI, body is divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area is assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. The total score ranges from 0 (no disease) to 72 (maximal disease)]; PGAPI ≤15 [using VAS on a scale of 0 (no pain) to (serious pain)]; PGADA ≤20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤0.5; LEI score ≤1 with participants with enthesitis at baseline.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.8] | 0 [0.0 to 5.6] | 0 [0.0 to 2.5]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.6] | 0 [0.0 to 5.6] | 10.5 [0.0 to 27.0]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 11.1 [0.0 to 28.4] | 5.3 [0.0 to 17.9] | 12.5 [0.0 to 41.7] | 5.3 [0.0 to 17.9]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 5.6 [0.0 to 18.9] | 10.5 [0.0 to 27.0] | 11.1 [0.0 to 37.2] | 0 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-9.9 to 20.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-5.3 to 5.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -5.3, 95% CI 2-sided [-27.6 to 17.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -10.5, 95% CI 2-sided [-29.6 to 8.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 5.8, 95% CI 2-sided [-17.2 to 28.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-19.5 to 19.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 5.6, 95% CI 2-sided [-10.3 to 21.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 10.5, 95% CI 2-sided [-8.4 to 29.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

5. Secondary Outcome: Change From Baseline in Disease Activity in Psoriatic Arthritis (DAPSA) at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. The DAPSA score has a lower bound of 0 and has no upper bound. A higher DAPSA score indicated more active disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 48.0 (25.55) | 30.3 (10.43) | 38.8 (20.82) | 33.8 (17.55)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -12.5 (11.96) | -5.3 (9.12) | -10.9 (8.39) | -7.5 (11.72)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -19.3 (14.30) | -9.4 (12.13) | -14.2 (10.45) | -6.5 (8.41)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -28.4 (15.67) | -12.4 (11.06) | -17.8 (12.96) | -10.6 (8.87)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -27.4 (17.09) | -18.0 (11.00) | -25.2 (16.60) | -9.3 (9.81)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -28.1 (13.42) | -17.4 (12.16) | -25.1 (14.55) | -11.3 (12.18)

6. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Psoriasis (PhGAP) at Weeks 2, 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the Body Surface Area (BSA) at Baseline
Description: The PhGAP is used to determine the participant's psoriasis lesions overall at a given time point. The participant's psoriasis disease activity is assessed by a physician according to the grades of induration, erythema, and scaling on a scale of 0 to 5. The sum of the three grades is used to obtain the total average score. PhGAP is based on the total average score on a scale of 0-5 where, 0 = cleared, 1 = minimal, 2 = mild, 3 = moderate, 4 = marked, and 5 = severe. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
score on a scale
  Baseline | 3 (1.2) | 2 (0.8) | 2 (0.5) | 2 (0.5)
  Change From Baseline at Week 2: number analyzed (Participants) | 8 | 5 | 4 | 3
  Change From Baseline at Week 2 | -1 (0.5) | 0 (0.0) | 0 (0.5) | 0 (0.0)
  Change From Baseline at Week 4 | -1 (1.0) | 0 (0.5) | -1 (1.0) | 0 (0.5)
  Change From Baseline at Week 8 | -1 (1.0) | -1 (0.7) | -1 (0.8) | -1 (1.0)
  Change From Baseline at Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Change From Baseline at Week 12 | -1 (1.3) | -1 (1.1) | -2 (0.6) | 0 (1.3)
  Change From Baseline at Week 16 | -1 (0.7) | -1 (0.8) | -2 (0.6) | -1 (1.4)

7. Secondary Outcome: Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) at Weeks 4, 8, 12, and 16 in Participants With Psoriatic Nail Involvement at Baseline
Description: mNAPSI is used to assess each nail abnormality for each of the participant's nails. Three features or groups of features (pitting, onycholysis together with oil-drop dyschromia, and crumbling) of each fingernail are graded on a scale from 0 (no onycholysis together with oil-drop dyschromia, no pitting, no crumbling) to 3 (>30 onycholysis together with oil-drop dyschromia, >50 pitting, >50% crumbling). Four features (leukonychia, splinter, hemorrhages, hyperkeratosis, and red spots in the lunula) are graded with the score of 1 = present or 0 = absent for each fingernail. Each finger has a score between 0 and 13. The total mNAPSI score is the sum of all abnormalities individual score across all fingers, and the total mNAPSI score ranges from 0 to 130. Lower numbers indicate fewer nail abnormalities. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriatic nail involvement at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 9 | 11 | 6 | 13
score on a scale
  Baseline | 19 (15.1) | 15 (12.9) | 24 (32.3) | 14 (12.9)
  Change From Baseline at Week 4: number analyzed (Participants) | 9 | 10 | 6 | 13
  Change From Baseline at Week 4 | -3 (3.5) | 1 (4.5) | -3 (10.0) | 0 (8.2)
  Change From Baseline at Week 8: number analyzed (Participants) | 9 | 11 | 6 | 12
  Change From Baseline at Week 8 | -3 (5.1) | -1 (5.9) | -6 (19.4) | -2 (5.0)
  Change From Baseline at Week 12: number analyzed (Participants) | 9 | 11 | 5 | 12
  Change From Baseline at Week 12 | -4 (6.0) | 0 (5.4) | -9 (23.2) | -3 (10.6)
  Change From Baseline at Week 16: number analyzed (Participants) | 8 | 11 | 6 | 13
  Change From Baseline at Week 16 | 0 (10.8) | -3 (9.6) | -14 (23.7) | -2 (9.2)

8. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) at Weeks 4, 8, 12, and 16 in Participants With Enthesitis at Baseline
Description: Enthesitis is assessed using LEI. The enthesitis examination by LEI evaluates the presence or absence of pain by applying local pressure on 6 anatomical sites: medial femoral condyle (left and right), lateral epicondyle (left and right), and the achilles tendon insertion (left and right). Enthesitis at each site is scored as 0 (enthesitis absent) and 1 (enthesitis present). LEI is derived as the sum of the enthesitis score over the 6 sites mentioned above. The total score ranges from 0 to 6, higher scores indicates greater degree of enthesitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 10 | 9 | 6 | 11
score on a scale
  Baseline | 2 (1.6) | 2 (1.4) | 2 (1.4) | 2 (1.7)
  Change From Baseline at Week 4 | -1 (0.8) | 0 (0.7) | -1 (1.1) | 0 (1.5)
  Change From Baseline at Week 8: number analyzed (Participants) | 10 | 9 | 6 | 10
  Change From Baseline at Week 8 | -1 (0.8) | -1 (1.2) | -2 (1.5) | 0 (1.3)
  Change From Baseline at Week 12: number analyzed (Participants) | 10 | 9 | 5 | 10
  Change From Baseline at Week 12 | -1 (1.4) | -1 (1.6) | -2 (1.8) | 0 (1.2)
  Change From Baseline at Week 16 | -1 (1.2) | -1 (1.5) | -2 (1.6) | 0 (1.5)

9. Secondary Outcome: Change From Baseline in 12-Item Psoriatic Arthritis Impact of Disease (PsAID-12) Score at Weeks 4 and 16
Description: The PsAID questionnaire assesses the impact of PsA on people's lives. The PsAID is calculated based on 12 numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. Total score is calculated as the sum of the individual scores, (some of which were multiplied by a weighting factor) divided by 20 for a total possible score of 0 to 10, where higher score indicates worse impact of disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 4.82 (1.857) | 4.46 (2.115) | 5.28 (1.765) | 4.44 (2.071)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -1.71 (1.282) | -1.39 (1.214) | -1.73 (1.645) | -0.10 (1.520)
  Change From Baseline at Week 16 | -2.06 (1.314) | -2.04 (1.740) | -2.56 (2.062) | -0.52 (2.176)

10. Secondary Outcome: Percentage of Participants With PASDAS Low Disease Activity (LDA) at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. It includes components of PGADA [using VAS on a scale of 0=very well to 100=very poor]; PhGADA [using VAS on a scale of 0=no disease activity to 100=maximum disease activity]; 36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains to determine a physical component summary (PCS) with a score range of 0-100, higher scores indicates better health status]; TJC68; SJC66; leeds enthesitis index(LEI) [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis]; Tender dactylitis count (TDC) [with a score range of 0 to 60, higher score indicates higher degree of dactylitis]; C-reactive protein (CRP). Total score is calculated as the sum of the individual scores (each score adjusted by weighting factors). The score of PASDAS ranges from 0 to 10, lower scores indicates better function. PASDAS LDA is defined as PASDAS ≤ 3.2.
Time Frame: Weeks 4, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Week 4 | 21.1 [0.1 to 42.0] | 11.1 [0.0 to 28.4] | 0 [0.0 to 6.3] | 5.0 [0.0 to 17.1]
  Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Week 16 | 38.9 [13.6 to 64.2] | 42.1 [17.3 to 66.9] | 50.0 [9.1 to 90.9] | 15.0 [0.0 to 33.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 16.1, 95% CI 2-sided [-9.7 to 41.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 6.1, 95% CI 2-sided [-16.5 to 28.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 23.9, 95% CI 2-sided [-8.8 to 56.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 27.1, 95% CI 2-sided [-5.2 to 59.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

11. Secondary Outcome: Percentage of Participants Who Achieved PASDAS Remission at Weeks 4 and 16
Description: PASDAS is a composite disease activity measure for psoriatic arthritis. It includes components of PGADA [using VAS on a scale of 0=very well to 100=very poor]; PhGADA [using VAS on a scale of 0=no disease activity to 100=maximum disease activity]; 36-item short form survey (SF-36) [a questionnaire which measures quality of life across eight domains to determine a physical component summary (PCS) with a score range of 0-100, higher scores indicates better health status];TJC68;SJC66; leeds enthesitis index(LEI) [assessed at 6 sites with a score range of 0 to 6, higher scores indicates higher degree of enthesitis]; Tender dactylitis count (TDC) [with a score range of 0 to 60, higher score indicates higher degree of dactylitis]; C-reactive protein (CRP). Total score is calculated as the sum of the individual scores (each score adjusted by weighting factors). The score of PASDAS ranges from 0 to 10, lower scores indicates better function. PASDAS remission is defined as PASDAS ≤ 1.9.
Time Frame: Weeks 4, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Week 4 | 0 [0.0 to 2.6] | 0 [0.0 to 2.8] | 0 [0.0 to 6.3] | 0 [0.0 to 2.5]
  Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Week 16 | 16.7 [0.0 to 36.7] | 10.5 [0.0 to 27.0] | 12.5 [0.0 to 41.7] | 5.0 [0.0 to 17.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-5.1 to 5.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-5.3 to 5.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 11.7, 95% CI 2-sided [-13.3 to 36.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 5.5, 95% CI 2-sided [-16.4 to 27.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

12. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 26.3 [3.9 to 48.7] | 5.6 [0.0 to 18.9] | 11.1 [0.0 to 37.2] | 10.5 [0.0 to 27.0]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 52.6 [27.5 to 77.7] | 27.8 [4.3 to 51.2] | 33.3 [0.0 to 69.7] | 10.0 [0.0 to 25.6]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 73.7 [51.3 to 96.1] | 36.8 [12.5 to 61.2] | 55.6 [17.5 to 93.6] | 31.6 [8.0 to 55.1]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 77.8 [55.8 to 99.8] | 63.2 [38.8 to 87.5] | 75.0 [38.7 to 100.0] | 42.1 [17.3 to 66.9]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 88.9 [71.6 to 100.0] | 52.6 [27.5 to 77.7] | 77.8 [45.1 to 100.0] | 45.0 [20.7 to 69.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.20, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 15.8, 95% CI 2-sided [-13.6 to 45.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.60, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = -5.0, 95% CI 2-sided [-27.8 to 17.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.008, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 42.6, 95% CI 2-sided [11.5 to 73.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.17, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 17.8, 95% CI 2-sided [-12.0 to 47.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.011, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 42.1, 95% CI 2-sided [8.1 to 76.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.69, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 5.3, 95% CI 2-sided [-30.1 to 40.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.033, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 35.7, 95% CI 2-sided [0.9 to 70.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.19, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 21.1, 95% CI 2-sided [-15.2 to 57.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 43.9, 95% CI 2-sided [12.4 to 75.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.63, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 7.6, 95% CI 2-sided [-28.8 to 44.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

13. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 50% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR50 response is achieved when the participant has: ≥ 50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.8] | 0 [0.0 to 5.6] | 5.3 [0.0 to 17.9]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 10.5 [0.0 to 27.0] | 5.6 [0.0 to 18.9] | 0 [0.0 to 5.6] | 5.0 [0.0 to 17.1]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 31.6 [8.0 to 55.1] | 26.3 [3.9 to 48.7] | 11.1 [0.0 to 37.2] | 10.5 [0.0 to 27.0]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 55.6 [29.8 to 81.3] | 42.1 [17.3 to 66.9] | 37.5 [0.0 to 77.3] | 10.5 [0.0 to 27.0]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 27.8 [4.3 to 51.2] | 47.4 [22.3 to 72.5] | 33.3 [0.0 to 69.7] | 15.0 [0.0 to 33.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.98, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 0.0, 95% CI 2-sided [-19.5 to 19.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.50, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = -5.3, 95% CI 2-sided [-20.7 to 10.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.54, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 5.5, 95% CI 2-sided [-16.4 to 27.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.92, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 0.6, 95% CI 2-sided [-19.0 to 20.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.13, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 21.1, 95% CI 2-sided [-9.3 to 51.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.22, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 15.8, 95% CI 2-sided [-13.6 to 45.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 45.0, 95% CI 2-sided [12.8 to 77.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.039, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 31.6, 95% CI 2-sided [0.2 to 63.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.34, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 12.8, 95% CI 2-sided [-18.4 to 44.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.040, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Difference in response rates = 32.4, 95% CI 2-sided [-0.1 to 64.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

14. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 70% Improvement Response at Weeks 2, 4, 8, 12, and 16
Description: ACR70 response is achieved when the participant has: ≥ 70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGADA using a VAS on a scale of 0 (very well) to 100 (very poor); PHGADA using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity); HAQ-DI inclusive of activities scored on a scale of 0 (no disability) to 3 (completely disabled); HAQ-DI pain assessment using VAS on a scale of 0 (no pain) to 100 (serious pain); and hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.8] | 0 [0.0 to 5.6] | 0 [0.0 to 2.6]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.8] | 0 [0.0 to 5.6] | 0 [0.0 to 2.5]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 15.8 [0.0 to 34.8] | 10.5 [0.0 to 27.0] | 0 [0.0 to 5.6] | 5.3 [0.0 to 17.9]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 27.8 [4.3 to 51.2] | 26.3 [3.9 to 48.7] | 12.5 [0.0 to 41.7] | 0 [0.0 to 2.6]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 22.2 [0.2 to 44.2] | 31.6 [8.0 to 55.1] | 22.2 [0.0 to 54.9] | 10.0 [0.0 to 25.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-10.0 to 20.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-5.4 to 5.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-9.9 to 20.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-5.3 to 5.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 10.5, 95% CI 2-sided [-14.0 to 35.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-17.1 to 27.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 27.8, 95% CI 2-sided [1.7 to 53.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 26.3, 95% CI 2-sided [1.3 to 51.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.2, 95% CI 2-sided [-16.3 to 40.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 21.6, 95% CI 2-sided [-8.2 to 51.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

15. Secondary Outcome: Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 2, 4, 8, 12, and 16
Description: TJC68 is an assessment of 68 joints. Each joint is evaluated as 'normal', 'tender', 'tender and swollen', or 'not able to evaluate'. It is derived as the sum of all tender joints. The overall tender joint count ranged from 0 to 68, with a higher score indicating a greater degree of tenderness. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
tender joint count
  Baseline | 22 (14.9) | 13 (8.5) | 17 (11.0) | 14 (11.6)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Change From Baseline at Week 2 | -6 (8.7) | -1 (5.2) | -5 (3.9) | -3 (6.6)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Change From Baseline at Week 4 | -9 (10.3) | -3 (7.9) | -7 (5.3) | -3 (4.6)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Change From Baseline at Week 8 | -13 (9.9) | -5 (6.3) | -7 (7.4) | -4 (4.8)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Change From Baseline at Week 12 | -13 (7.4) | -7 (7.4) | -10 (8.5) | -4 (4.5)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Change From Baseline at Week 16 | -14 (7.7) | -7 (7.9) | -10 (6.1) | -5 (8.3)

16. Secondary Outcome: Change From Baseline in ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 2, 4, 8, 12, and 16
Description: SJC66 is an assessment of 66 joints. Each joint was evaluated as 'normal', 'swollen', 'tender and swollen', or 'not able to evaluate'. It is derived as the sum of all swollen joints. The overall swollen joint count ranged from 0 to 66, with a higher score indicating a greater degree of swelling. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
swollen joint count
  Baseline | 14 (10.3) | 7 (3.3) | 11 (7.3) | 8 (5.9)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Change From Baseline at Week 2 | -3 (3.8) | -1 (3.5) | -5 (5.2) | -2 (4.7)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Change From Baseline at Week 4 | -5 (6.2) | -2 (2.9) | -4 (7.0) | -2 (3.1)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Change From Baseline at Week 8 | -9 (7.0) | -3 (4.0) | -6 (6.1) | -3 (2.9)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Change From Baseline at Week 12 | -8 (8.9) | -4 (3.1) | -8 (7.3) | -4 (2.9)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Change From Baseline at Week 16 | -8 (7.9) | -4 (3.8) | -8 (6.7) | -4 (3.9)

17. Secondary Outcome: Change From Baseline in Individual ACR Component: Patient's Global Assessment of Disease Activity (PGADA) at Weeks 2, 4, 8, 12, and 16
Description: PGADA is assessed by the participants using a VAS on a scale of 0 (very well) to 100 (very poor). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 54 (26.0) | 58 (22.8) | 47 (24.2) | 52 (24.0)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -15 (17.8) | -17 (26.6) | 3 (8.6) | -10 (12.6)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -23 (20.3) | -23 (32.2) | -3 (11.4) | -4 (16.6)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -24 (22.6) | -28 (33.8) | -4 (17.1) | -16 (23.4)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -27 (25.9) | -38 (29.9) | -29 (19.7) | -9 (24.7)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -31 (26.4) | -34 (28.5) | -25 (25.3) | -12 (23.5)

18. Secondary Outcome: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PhGADA) at Weeks 2, 4, 8, 12, and 16
Description: PhGADA is assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 68 (16.4) | 56 (14.3) | 65 (13.1) | 62 (13.4)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -17 (12.3) | -4 (11.0) | -12 (9.2) | -8 (9.8)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -23 (14.5) | -12 (18.6) | -29 (14.8) | -8 (11.5)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -35 (15.1) | -17 (17.4) | -35 (13.6) | -21 (13.7)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -36 (18.8) | -26 (22.4) | -42 (20.8) | -21 (21.8)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -37 (16.4) | -27 (21.6) | -44 (21.0) | -19 (20.2)

19. Secondary Outcome: Change From Baseline in Individual ACR Component: Health Assessment Questionnaire Disability Index (HAQ-DI)'s Pain Assessment at Weeks 2, 4, 8, 12, and 16
Description: HAQ-DI's pain assessment is done using VAS on a scale of 0 (no pain) to 100 (serious pain). A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 60 (24.7) | 45 (22.3) | 48 (24.3) | 56 (24.2)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -16 (15.2) | -4 (16.7) | -5 (9.5) | -8 (11.5)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -24 (20.9) | -13 (18.6) | -10 (9.8) | -1 (14.3)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -33 (20.9) | -13 (23.4) | -3 (17.3) | -11 (25.3)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -33 (23.7) | -19 (21.0) | -28 (20.7) | -8 (23.3)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -29 (24.5) | -17 (26.5) | -27 (15.2) | -12 (21.7)

20. Secondary Outcome: Change From Baseline in Individual ACR Component: High-Sensitivity C-Reactive Protein (hsCRP) at Weeks 2, 4, 8, 12, and 16
Description: The hsCRP is the ACR core set measure of acute phase reactant. It was measured at the central laboratory to help assess the effect of filgotinib on the participant's psoriatic arthritis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
mg/L
  Baseline | 8.08 (9.335) | 3.14 (2.673) | 10.56 (16.354) | 7.11 (9.727)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Change From Baseline at Week 2 | -6.37 (8.518) | -0.10 (5.313) | -7.70 (11.874) | 0.50 (4.063)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Change From Baseline at Week 4 | -6.68 (8.998) | -0.95 (2.564) | -5.99 (8.981) | 3.96 (13.594)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Change From Baseline at Week 8 | -5.13 (11.271) | -0.69 (4.474) | -6.40 (9.740) | -1.15 (4.979)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Change From Baseline at Week 12 | -6.04 (8.518) | -1.11 (3.161) | -3.80 (7.334) | 2.25 (7.788)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Change From Baseline at Week 16 | -5.88 (9.195) | -0.47 (5.496) | -6.80 (10.918) | 1.05 (5.623)

21. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) C-Reactive Protein (CRP) at Weeks 2, 4, 8, 12, and 16
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA [using a VAS on a scale of 0 (very well) to 100 (very poor)] and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 4.9 (1.27) | 4.2 (0.78) | 4.5 (0.97) | 4.4 (0.92)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -0.9 (0.62) | -0.5 (0.74) | -0.9 (0.70) | -0.6 (0.83)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -1.2 (0.63) | -0.9 (1.04) | -1.2 (0.60) | -0.5 (0.65)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -1.8 (0.87) | -1.2 (0.71) | -1.2 (0.83) | -1.0 (0.66)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -1.9 (0.96) | -1.5 (0.89) | -1.9 (0.88) | -0.8 (0.78)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -1.8 (0.62) | -1.8 (0.97) | -2.0 (0.71) | -0.8 (0.92)

22. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) LDA at Weeks 2, 4, 8, 12, and 16
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) LDA is defined as DAS28(CRP) ≤ 3.2.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 31.6 [8.0 to 55.1] | 33.3 [8.8 to 57.9] | 33.3 [0.0 to 69.7] | 42.1 [17.3 to 66.9]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 36.8 [12.5 to 61.2] | 44.4 [18.7 to 70.2] | 55.6 [17.5 to 93.6] | 25.0 [3.5 to 46.5]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 63.2 [38.8 to 87.5] | 63.2 [38.8 to 87.5] | 33.3 [0.0 to 69.7] | 52.6 [27.5 to 77.7]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 66.7 [42.1 to 91.2] | 68.4 [44.9 to 92.0] | 62.5 [22.7 to 100.0] | 36.8 [12.5 to 61.2]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 50.0 [24.1 to 75.9] | 84.2 [65.2 to 100.0] | 66.7 [30.3 to 100.0] | 45.0 [20.7 to 69.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -10.5, 95% CI 2-sided [-46.3 to 25.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -8.8, 95% CI 2-sided [-45.3 to 27.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 11.8, 95% CI 2-sided [-22.1 to 45.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 19.4, 95% CI 2-sided [-15.6 to 54.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 10.5, 95% CI 2-sided [-26.0 to 47.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 10.5, 95% CI 2-sided [-26.0 to 47.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 29.8, 95% CI 2-sided [-6.3 to 66.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 31.6, 95% CI 2-sided [-3.8 to 67.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 5.0, 95% CI 2-sided [-32.0 to 42.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 39.2, 95% CI 2-sided [6.8 to 71.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

23. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) Remission at Weeks 2, 4, 8, 12, and 16
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the tender joint count (28 joints), swollen joint count (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) remission is defined as DAS28 (CRP) < 2.6.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 10.5 [0.0 to 27.0] | 11.1 [0.0 to 28.4] | 22.2 [0.0 to 54.9] | 10.5 [0.0 to 27.0]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 10.5 [0.0 to 27.0] | 27.8 [4.3 to 51.2] | 22.2 [0.0 to 54.9] | 15.0 [0.0 to 33.1]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 47.4 [22.3 to 72.5] | 26.3 [3.9 to 48.7] | 22.2 [0.0 to 54.9] | 26.3 [3.9 to 48.7]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 55.6 [29.8 to 81.3] | 42.1 [17.3 to 66.9] | 50.0 [9.1 to 90.9] | 21.1 [0.1 to 42.0]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 44.4 [18.7 to 70.2] | 52.6 [27.5 to 77.7] | 44.4 [6.4 to 82.5] | 20.0 [0.0 to 40.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-24.8 to 24.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.6, 95% CI 2-sided [-24.9 to 26.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = -4.5, 95% CI 2-sided [-30.5 to 21.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 12.8, 95% CI 2-sided [-18.4 to 44.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 21.1, 95% CI 2-sided [-14.1 to 56.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-33.3 to 33.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 34.5, 95% CI 2-sided [-0.3 to 69.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 21.1, 95% CI 2-sided [-13.0 to 55.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 24.4, 95% CI 2-sided [-9.7 to 58.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 32.6, 95% CI 2-sided [-1.0 to 66.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

24. Secondary Outcome: Time to Achieve DAS28 (CRP) LDA
Description: The DAS28 (CRP) is a measure of the participant's disease activity calculated using the TJC (28 joints), SJC (28 joints), PGADA (VAS; 0 = very well to 100 = very poor), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. DAS28 (CRP) LDA is defined as DAS28 (CRP) ≤ 3.2. Time to achieve DAS28 (CRP) LDA is the number of days from the first dose date of study drug administration to the first time when a participant achieves DAS28 (CRP) LDA.
Time Frame: Up to 19 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 18 | 17 | 7 | 17
days | 57 [17 to NA] — Upper bound of 95% CI was not estimable due to low number of participants with DAS28 (CRP) LDA. | 58 [16 to 113] | 29 [14 to 127] | 59 [15 to NA] — Upper bound of 95% CI was not estimable due to low number of participants with DAS28 (CRP) LDA.

25. Secondary Outcome: Percentage of Participants Who Achieved DAPSA LDA at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. The DAPSA score has a lower bound of 0 and has no upper bound. A higher DAPSA score indicated more active disease activity. DAPSA LDA is defined as DAPSA ≤ 14.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 15.8 [0.0 to 34.8] | 11.1 [0.0 to 28.4] | 22.2 [0.0 to 54.9] | 31.6 [8.0 to 55.1]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 31.6 [8.0 to 55.1] | 38.9 [13.6 to 64.2] | 44.4 [6.4 to 82.5] | 25.0 [3.5 to 46.5]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 52.6 [27.5 to 77.7] | 42.1 [17.3 to 66.9] | 33.3 [0.0 to 69.7] | 36.8 [12.5 to 61.2]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 61.1 [35.8 to 86.4] | 57.9 [33.1 to 82.7] | 62.5 [22.7 to 100.0] | 36.8 [12.5 to 61.2]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 44.4 [18.7 to 70.2] | 63.2 [38.8 to 87.5] | 55.6 [17.5 to 93.6] | 40.0 [16.0 to 64.0]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -15.8, 95% CI 2-sided [-47.6 to 16.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -20.5, 95% CI 2-sided [-51.3 to 10.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 6.6, 95% CI 2-sided [-26.8 to 39.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 13.9, 95% CI 2-sided [-20.8 to 48.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 15.8, 95% CI 2-sided [-20.7 to 52.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 5.3, 95% CI 2-sided [-31.0 to 41.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 24.3, 95% CI 2-sided [-12.4 to 60.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 21.1, 95% CI 2-sided [-15.2 to 57.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 4.4, 95% CI 2-sided [-32.3 to 41.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 23.2, 95% CI 2-sided [-12.5 to 58.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

26. Secondary Outcome: Percentage of Participants Who Achieved DAPSA Remission at Weeks 2, 4, 8, 12, and 16
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. The DAPSA score has a lower bound of 0 and has no upper bound. A higher DAPSA score indicated more active disease activity. DAPSA remission is defined as DAPSA ≤ 4.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 5.3 [0.0 to 17.9] | 0 [0.0 to 2.8] | 0 [0.0 to 5.6] | 5.3 [0.0 to 17.9]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 5.3 [0.0 to 17.9] | 5.6 [0.0 to 18.9] | 0 [0.0 to 5.6] | 5.0 [0.0 to 17.1]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 10.5 [0.0 to 27.0] | 5.3 [0.0 to 17.9] | 0 [0.0 to 5.6] | 10.5 [0.0 to 27.0]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 22.2 [0.2 to 44.2] | 31.6 [8.0 to 55.1] | 12.5 [0.0 to 41.7] | 5.3 [0.0 to 17.9]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 16.7 [0.0 to 36.7] | 21.1 [0.1 to 42.0] | 22.2 [0.0 to 54.9] | 10.0 [0.0 to 25.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-19.5 to 19.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -5.3, 95% CI 2-sided [-20.7 to 10.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.3, 95% CI 2-sided [-18.7 to 19.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.6, 95% CI 2-sided [-19.0 to 20.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-24.8 to 24.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -5.3, 95% CI 2-sided [-27.6 to 17.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 17.0, 95% CI 2-sided [-10.1 to 44.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 26.3, 95% CI 2-sided [-2.1 to 54.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 6.7, 95% CI 2-sided [-20.3 to 33.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 11.1, 95% CI 2-sided [-16.6 to 38.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

27. Secondary Outcome: Time to Achieve DAPSA LDA
Description: DAPSA is calculated by summing the following components: TJC68; SJC66; PGADA [using VAS on a scale of 0 (very well) to 100 very poor)]; PGAPI [using a VAS on a scale of 0 (no pain) to 100 (serious pain)] and CRP. DAPSA scores 0-4 = remission, 5-14 = low disease activity, 15-28 = moderate disease activity, and >28 = high disease activity. The DAPSA score has a lower bound of 0 and has no upper bound. A higher DAPSA score indicated more active disease activity. Time to achieve DAPSA LDA is the number of days from the first dose date of study drug administration to the first time when a participant achieves DAPSA LDA. If the DAPSA LDA is not achieved during main study phase, the time to achieve DAPSA LDA will be censored at the last non-missing DAPSA LDA assessment date during main study phase. If the component scores of DAPSA LDA are at different dates for a visit, the latest date will be used for the derivation of time to achieve DAPSA LDA.
Time Frame: Up to 19 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 18 | 18 | 7 | 18
days | 73 [31 to NA] — Upper bound of 95% CI was not estimable due to the low number of participants with DAPSA LDA. | 82 [29 to NA] — Upper bound of 95% CI was not estimable due to the low number of participants with DAPSA LDA. | 83 [15 to 127] | NA [16 to NA] — Median and Upper bound of 95% CI were not estimable due to the low number of participants with DAPSA LDA.

28. Secondary Outcome: Percentage of Participants Who Achieved Psoriatic Arthritis Response Criteria (PsARC) Response at Weeks 2, 4, 8, 12, and 16
Description: The PsARC response is defined as improvement in at least 2 of the following 4 criteria; ≥ 30% decrease in SJC66, ≥ 30% decrease in TJC68, ≥ 20% decrease in PGADA (VAS; 0 = very well to 100 = very poor), ≥ 20% decrease in PhGADA (VAS; 0 = no disease activity to 100 = maximum disease activity), and with at least one of the 2 joint criteria, with no deterioration in any other criteria.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: Participants in the FAS with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 9 | 20
percentage of participants
  Week 2: number analyzed (Participants) | 19 | 18 | 9 | 19
  Week 2 | 31.6 [8.0 to 55.1] | 16.7 [0.0 to 36.7] | 11.1 [0.0 to 37.2] | 31.6 [8.0 to 55.1]
  Week 4: number analyzed (Participants) | 19 | 18 | 9 | 20
  Week 4 | 57.9 [33.1 to 82.7] | 38.9 [13.6 to 64.2] | 44.4 [6.4 to 82.5] | 30.0 [7.4 to 52.6]
  Week 8: number analyzed (Participants) | 19 | 19 | 9 | 19
  Week 8 | 78.9 [58.0 to 99.9] | 47.4 [22.3 to 72.5] | 44.4 [6.4 to 82.5] | 57.9 [33.1 to 82.7]
  Week 12: number analyzed (Participants) | 18 | 19 | 8 | 19
  Week 12 | 72.2 [48.8 to 95.7] | 68.4 [44.9 to 92.0] | 75.0 [38.7 to 100.0] | 47.4 [22.3 to 72.5]
  Week 16: number analyzed (Participants) | 18 | 19 | 9 | 20
  Week 16 | 88.9 [71.6 to 100.0] | 57.9 [33.1 to 82.7] | 77.8 [45.1 to 100.0] | 45.0 [20.7 to 69.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-34.8 to 34.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; Difference in response rates = -14.9, 95% CI 2-sided [-47.4 to 17.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 27.9, 95% CI 2-sided [-7.2 to 63.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 8.9, 95% CI 2-sided [-26.6 to 44.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 21.1, 95% CI 2-sided [-13.0 to 55.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -10.5, 95% CI 2-sided [-47.4 to 26.3] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 24.9, 95% CI 2-sided [-11.1 to 60.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 21.1, 95% CI 2-sided [-14.9 to 57.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 43.9, 95% CI 2-sided [12.4 to 75.4] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.9, 95% CI 2-sided [-23.4 to 49.1] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

29. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, where 0 = none, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A higher score indicates more severe disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
score on a scale
  Baseline | 9.5 (6.70) | 13.8 (14.12) | 6.5 (5.90) | 9.6 (10.60)
  Change From Baseline at Week 4 | -2.2 (5.19) | -5.0 (5.14) | -1.8 (1.54) | -1.1 (5.41)
  Change From Baseline at Week 8 | -3.4 (4.91) | -5.5 (4.93) | -3.0 (1.98) | -5.6 (7.03)
  Change From Baseline at Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Change From Baseline at Week 12 | -3.7 (5.65) | -5.6 (6.13) | -3.0 (2.10) | -4.9 (7.12)
  Change From Baseline at Week 16 | -5.5 (7.80) | -7.0 (7.69) | -5.2 (4.56) | -6.4 (9.85)

30. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 50% Improvement (PASI50) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI50, the improvement threshold from baseline in PASI score is 50%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
percentage of participants
  Week 4 | 37.5 [0.0 to 77.3] | 40.0 [0.0 to 92.9] | 50.0 [0.0 to 100.0] | 0 [0.0 to 12.5]
  Week 8 | 25.0 [0.0 to 61.3] | 40.0 [0.0 to 92.9] | 50.0 [0.0 to 100.0] | 50.0 [0.0 to 100.0]
  Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Week 12 | 57.1 [13.3 to 100.0] | 40.0 [0.0 to 92.9] | 100.0 [83.3 to 100.0] | 50.0 [0.0 to 100.0]
  Week 16 | 62.5 [22.7 to 100.0] | 40.0 [0.0 to 92.9] | 100.0 [87.5 to 100.0] | 25.0 [0.0 to 79.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 37.5, 95% CI 2-sided [-14.8 to 89.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 40.0, 95% CI 2-sided [-25.4 to 100.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -25.0, 95% CI 2-sided [-100.0 to 51.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = -10.0, 95% CI 2-sided [-97.7 to 77.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 7.1, 95% CI 2-sided [-73.7 to 88.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = -10.0, 95% CI 2-sided [-97.7 to 77.7] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 37.5, 95% CI 2-sided [-35.3 to 100.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 15.0, 95% CI 2-sided [-67.9 to 97.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

31. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 75% Improvement (PASI75) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI75, the improvement threshold from baseline in PASI score is 75%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
percentage of participants
  Week 4 | 12.5 [0.0 to 41.7] | 20.0 [0.0 to 65.1] | 0 [0.0 to 12.5] | 0 [0.0 to 12.5]
  Week 8 | 25.0 [0.0 to 61.3] | 40.0 [0.0 to 92.9] | 25.0 [0.0 to 79.9] | 0 [0.0 to 12.5]
  Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Week 12 | 42.9 [0.0 to 86.7] | 40.0 [0.0 to 92.9] | 66.7 [0.0 to 100.0] | 0 [0.0 to 12.5]
  Week 16 | 62.5 [22.7 to 100.0] | 20.0 [0.0 to 65.1] | 75.0 [20.1 to 100.0] | 25.0 [0.0 to 79.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 12.5, 95% CI 2-sided [-29.2 to 54.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 20.0, 95% CI 2-sided [-37.6 to 77.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 25.0, 95% CI 2-sided [-23.8 to 73.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 40.0, 95% CI 2-sided [-25.4 to 100.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 42.9, 95% CI 2-sided [-13.4 to 99.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 40.0, 95% CI 2-sided [-25.4 to 100.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 37.5, 95% CI 2-sided [-35.3 to 100.0] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = -5.0, 95% CI 2-sided [-82.5 to 72.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

32. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 90% Improvement (PASI90) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI90, the improvement threshold from baseline in PASI score is 90%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
percentage of participants
  Week 4 | 0 [0.0 to 6.3] | 0 [0.0 to 10.0] | 0 [0.0 to 12.5] | 0 [0.0 to 12.5]
  Week 8 | 12.5 [0.0 to 41.7] | 0 [0.0 to 10.0] | 25.0 [0.0 to 79.9] | 0 [0.0 to 12.5]
  Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Week 12 | 14.3 [0.0 to 47.4] | 20.0 [0.0 to 65.1] | 66.7 [0.0 to 100.0] | 0 [0.0 to 12.5]
  Week 16 | 25.0 [0.0 to 61.3] | 20.0 [0.0 to 65.1] | 50.0 [0.0 to 100.0] | 0 [0.0 to 12.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-18.8 to 18.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.5 to 22.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 12.5, 95% CI 2-sided [-29.2 to 54.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.5 to 22.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 14.3, 95% CI 2-sided [-31.3 to 59.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 20.0, 95% CI 2-sided [-37.6 to 77.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 25.0, 95% CI 2-sided [-23.8 to 73.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 20.0, 95% CI 2-sided [-37.6 to 77.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

33. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 100% Improvement (PASI100) Response at Weeks 4, 8, 12, and 16 in Participants With Psoriasis Covering ≥ 3% of the BSA at Baseline
Description: PASI is assessed in participants with psoriasis covering ≥ 3% of the BSA at Baseline. PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head and neck, trunk, upper limbs, and lower limbs. Each of these areas are assessed separately for the percentage of the area involved and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement). The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). For PASI100, the improvement threshold from baseline in PASI score is 100%. A higher score indicates more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: Participants in the FAS with psoriasis covering ≥ 3% of the BSA at baseline and with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 8 | 5 | 4 | 4
percentage of participants
  Week 4 | 0 [0.0 to 6.3] | 0 [0.0 to 10.0] | 0 [0.0 to 12.5] | 0 [0.0 to 12.5]
  Week 8 | 0 [0.0 to 6.3] | 0 [0.0 to 10.0] | 25.0 [0.0 to 79.9] | 0 [0.0 to 12.5]
  Week 12: number analyzed (Participants) | 7 | 5 | 3 | 4
  Week 12 | 14.3 [0.0 to 47.4] | 0 [0.0 to 10.0] | 66.7 [0.0 to 100.0] | 0 [0.0 to 12.5]
  Week 16 | 12.5 [0.0 to 41.7] | 20.0 [0.0 to 65.1] | 25.0 [0.0 to 79.9] | 0 [0.0 to 12.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-18.8 to 18.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.5 to 22.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-18.8 to 18.8] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.5 to 22.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 14.3, 95% CI 2-sided [-31.3 to 59.9] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; Difference in response rates = 0.0, 95% CI 2-sided [-22.5 to 22.5] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 12.5, 95% CI 2-sided [-29.2 to 54.2] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; Difference in response rates = 20.0, 95% CI 2-sided [-37.6 to 77.6] — 95% CI for difference in response rates were based on normal approximation method with a continuity correction

34. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index at Weeks 4, 8, 12, and 16 in Participants With Enthesitis at Baseline
Description: The enthesitis examination is based on the 16 anatomical sites: the medial epicondyle (left and right), the lateral epicondyle (left and right), the supraspinatus insertion (left and right), the bilateral greater trochanter (left and right), the quadriceps tendon insertion into superior border of patella (left and right), the patellar ligament insertion into inferior pole of patella or tibial tuberosity (left and right), the achilles tendon insertion (left and right), and the plantar fascia insertion (left and right). Enthesitis at each site is scored as either 0 (enthesitis absent) and 1 (enthesitis present). SPARCC enthesitis index has an overall total score ranging from 0 to 16. Higher score indicates a greater number of sites that are affected by enthesitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with enthesitis at baseline and with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 10 | 9 | 6 | 11
score on a scale
  Baseline | 4 (3.4) | 4 (2.4) | 4 (1.7) | 5 (4.5)
  Change From Baseline at Week 4 | -2 (2.6) | 0 (2.0) | -2 (1.2) | 0 (3.1)
  Change From Baseline at Week 8: number analyzed (Participants) | 10 | 9 | 6 | 10
  Change From Baseline at Week 8 | -2 (2.4) | -1 (1.6) | -3 (1.9) | -2 (3.3)
  Change From Baseline at Week 12: number analyzed (Participants) | 10 | 9 | 5 | 10
  Change From Baseline at Week 12 | -3 (3.5) | -2 (1.8) | -2 (1.5) | -1 (1.7)
  Change From Baseline at Week 16 | -3 (3.3) | -2 (2.6) | -3 (1.5) | -1 (3.2)

35. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI) at Weeks 4, 8, 12, and 16 in Participants With Dactylitis at Baseline
Description: LDI quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with an at least 10% difference in the ratio of circumference of the affected digit to the contralateral digit (digit on opposite hand or foot), or if contralateral digit is also affected, values from a standard reference table. Total score= {{[Circumference involved digit/ Circumference contralateral Digit (or Tables)] - 1}x 100} x Tenderness score. Tenderness score (0 = no tenderness, and 1 = tender). The difference between circumference of affected finger and contralateral not affected digit cannot be defined for maximum value. Therefore, it is difficult to provide scale range for the final score. No theoretical range exists for the Leeds Dactylitis Index. Lower Leeds Dactylitis Index score represent better outcome. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with dactylitis at baseline were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 6 | 3 | 1 | 5
score on a scale
  Baseline | 69.5 (56.62) | 28.9 (17.35) | 159.1 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. | 15.2 (19.45)
  Change From Baseline at Week 4 | -13.4 (16.81) | 13.0 (19.44) | -159.1 (NA) — SD cannot be calculated for 1 participant. | 13.3 (30.64)
  Change From Baseline at Week 8 | -40.8 (45.15) | -2.5 (18.34) | -159.1 (NA) — SD cannot be calculated for 1 participant. | 3.6 (40.81)
  Change From Baseline at Week 12 | -49.3 (40.86) | -14.0 (9.80) | -159.1 (NA) — SD cannot be calculated for 1 participant. | 2.1 (44.13)
  Change From Baseline at Week 16 | -40.2 (51.12) | 8.4 (41.91) | -159.1 (NA) — SD cannot be calculated for 1 participant. | 2.0 (31.30)

36. Secondary Outcome: Change From Baseline in Tender Dactylitis Count (TDC) at Weeks 4, 8, 12, and 16 in Participants With Dactylitis at Baseline
Description: Tender score (0 = no tenderness, 1 = tender, 2 = tender and wince, 3 = tender and withdraw) is collected for Dactylitis Assessments on the Dactylitis Score Sheet that is used for calculation of LDI total score. Tender dactylitis count (TDC) equals the number of tender fingers and toes (tendor score >0). For participants with dactylitis status absent for all the fingers and toes, the TDC is set as 0. The total score range of TDC is from 0 to 60, higher scores indicate greater presence of dactylitis. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with dactylitis at baseline were analyzed.
Measure: Mean (Standard Deviation); unit: tender dactylitis count
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 6 | 3 | 1 | 5
tender dactylitis count
  Baseline | 4 (4.1) | 2 (1.0) | 6 (NA) — SD cannot be calculated for 1 participant. | 1 (1.3)
  Change From Baseline at Week 4 | -1 (0.9) | 1 (1.0) | -6 (NA) — SD cannot be calculated for 1 participant. | 0 (1.5)
  Change From Baseline at Week 8 | -3 (3.3) | 0 (1.5) | -6 (NA) — SD cannot be calculated for 1 participant. | 0 (2.1)
  Change From Baseline at Week 12 | -3 (3.0) | -1 (1.5) | -6 (NA) — SD cannot be calculated for 1 participant. | 0 (2.2)
  Change From Baseline at Week 16 | -3 (3.3) | 0 (2.1) | -6 (NA) — SD cannot be calculated for 1 participant. | 0 (1.5)

37. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Weeks 2, 4, 8, 12, and 16
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). When 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing. A negative change from baseline indicates improvement (less disability).
Time Frame: Baseline, 2, 4, 8, 12, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 1.05 (0.601) | 0.80 (0.547) | 0.95 (0.630) | 0.92 (0.602)
  Change From Baseline at Week 2: number analyzed (Participants) | 19 | 18 | 8 | 19
  Change From Baseline at Week 2 | -0.13 (0.293) | -0.09 (0.345) | 0.03 (0.332) | -0.08 (0.321)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | -0.20 (0.264) | -0.24 (0.474) | -0.16 (0.297) | -0.01 (0.337)
  Change From Baseline at Week 8: number analyzed (Participants) | 19 | 19 | 8 | 19
  Change From Baseline at Week 8 | -0.37 (0.387) | -0.24 (0.516) | -0.16 (0.281) | -0.12 (0.407)
  Change From Baseline at Week 12: number analyzed (Participants) | 18 | 19 | 7 | 19
  Change From Baseline at Week 12 | -0.33 (0.374) | -0.20 (0.477) | -0.39 (0.274) | -0.07 (0.438)
  Change From Baseline at Week 16: number analyzed (Participants) | 18 | 19 | 8 | 20
  Change From Baseline at Week 16 | -0.33 (0.407) | -0.33 (0.575) | -0.34 (0.297) | -0.19 (0.487)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.94, MMRM — P-value was calculated from mixed-effects model for repeated measures (MMRM) including treatment, visit (categorical), treatment by visit, stratification factors, baseline value as fixed effects, and participants being the random effect; LS Mean Treatment Difference = -0.01, 95% CI 2-sided [-0.22 to 0.20], Standard Error of Mean 0.104
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 2; Test type: Superiority; p = 0.81, MMRM — P-value was calculated from MMRM including treatment, visit (categorical), treatment by visit, stratification factors, baseline value as fixed effects, and participants being the random effect; LS Mean Treatment Difference = 0.03, 95% CI 2-sided [-0.18 to 0.24], Standard Error of Mean 0.105
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.13, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.17, 95% CI 2-sided [-0.39 to 0.05], Standard Error of Mean 0.112
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.073, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.21, 95% CI 2-sided [-0.43 to 0.02], Standard Error of Mean 0.113
Statistical Analysis 5: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.083, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.22, 95% CI 2-sided [-0.46 to 0.03], Standard Error of Mean 0.124
Statistical Analysis 6: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 8; Test type: Superiority; p = 0.28, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.14, 95% CI 2-sided [-0.38 to 0.11], Standard Error of Mean 0.124
Statistical Analysis 7: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.038, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.28, 95% CI 2-sided [-0.54 to -0.02], Standard Error of Mean 0.130
Statistical Analysis 8: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 12; Test type: Superiority; p = 0.25, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.15, 95% CI 2-sided [-0.41 to 0.11], Standard Error of Mean 0.129
Statistical Analysis 9: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.41, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.11, 95% CI 2-sided [-0.39 to 0.16], Standard Error of Mean 0.139
Statistical Analysis 10: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.26, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = -0.16, 95% CI 2-sided [-0.43 to 0.12], Standard Error of Mean 0.138

38. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) Score at Weeks 4 and 16
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Higher scores indicate less fatigue. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 32.5 (9.83) | 33.9 (13.06) | 33.4 (10.66) | 31.4 (10.37)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | 4.6 (9.75) | 4.1 (8.53) | 0.5 (7.23) | 1.6 (6.53)
  Change From Baseline at Week 16 | 5.6 (9.45) | 6.4 (10.42) | 4.6 (9.18) | 2.4 (9.27)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.14, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 3.4, 95% CI 2-sided [-1.1 to 7.9], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.18, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 3.1, 95% CI 2-sided [-1.5 to 7.7], Standard Error of Mean 2.30
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.15, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 3.7, 95% CI 2-sided [-1.4 to 8.7], Standard Error of Mean 2.53
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.062, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 4.8, 95% CI 2-sided [-0.3 to 9.9], Standard Error of Mean 2.54

39. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) of the 36-Item Short-Form Version 2 (SF-36v2) at Weeks 4 and 16
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). MCS consists of social functioning, vitality, mental health, and role-emotional scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. A positive change from baseline indicated improvement (better health status).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 200 mg (Main Study): Participants will receive filgotinib 200 mg orally once daily + placebo to match (PTM) filgotinib 100 mg orally once daily + PTM adalimumab injection every two weeks for 16 weeks.
- Filgotinib 100 mg (Main Study): Participants will receive PTM filgotinib 200 mg orally one daily + filgotinib 100 mg orally once daily + PTM adalimumab every two weeks for 16 weeks.
- Adalimumab (Main Study): Participants will receive PTM filgotinib 200 mg orally once daily + PTM filgotinib 100 mg orally once daily + adalimumab 40 mg injection every two weeks for 16 weeks.
- Placebo (Main Study): Participants will receive PTM filgotinib 200 mg orally once daily + PTM filgotinib 100 mg orally once daily + PTM adalimumab injection every two weeks for 16 weeks.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 49.9 (12.48) | 50.5 (11.43) | 44.8 (7.67) | 48.9 (9.27)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | 3.3 (9.66) | 0.4 (9.40) | 0.6 (6.80) | -0.4 (5.58)
  Change From Baseline at Week 16 | 2.8 (10.34) | 0.2 (9.42) | 2.9 (9.31) | 0.3 (5.95)

40. Secondary Outcome: Change From Baseline in Physical Component Score (PCS) of the SF-36v2 at Weeks 4 and 16
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). PCS consists of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. A positive change from baseline indicates improvement (better health status).
Time Frame: Baseline, 4, and 16 weeks
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Filgotinib 100 mg (Main Study): Participants will receive PTM filgotinib 200 mg orally once daily + filgotinib 100 mg orally once daily + PTM adalimumab every two weeks for 16 weeks.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 19 | 19 | 8 | 20
score on a scale
  Baseline | 37.1 (8.11) | 39.2 (9.60) | 39.2 (7.58) | 37.2 (7.83)
  Change From Baseline at Week 4: number analyzed (Participants) | 19 | 18 | 8 | 20
  Change From Baseline at Week 4 | 6.4 (5.87) | 5.6 (7.00) | 2.9 (7.12) | 1.1 (5.24)
  Change From Baseline at Week 16 | 8.4 (6.86) | 7.4 (9.80) | 8.1 (7.73) | 4.6 (7.85)
Statistical Analysis 1: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 5.3, 95% CI 2-sided [1.9 to 8.6], Standard Error of Mean 1.68
Statistical Analysis 2: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 4; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 4.9, 95% CI 2-sided [1.5 to 8.3], Standard Error of Mean 1.71
Statistical Analysis 3: Comparison: Filgotinib 200 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.076, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 3.8, 95% CI 2-sided [-0.4 to 8.0], Standard Error of Mean 2.09
Statistical Analysis 4: Comparison: Filgotinib 100 mg (Main Study) vs Placebo (Main Study); Week 16; Test type: Superiority; p = 0.10, MMRM — [p-value comment as in outcome 37, analysis 2]; LS Mean Treatment Difference = 3.5, 95% CI 2-sided [-0.7 to 7.7], Standard Error of Mean 2.10

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 50 weeks plus 30 days; All-Cause Mortality: Randomization up to 50 weeks plus 30 days
Description: Adverse Events: Safety Analysis Set included all participants who took at least 1 dose of study drug. All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Groups:
- Filgotinib 200 mg From Filgotinib 200 mg (LTE): Filgotinib 200 mg tablet orally once daily + PTM filgotinib 100 mg tablet orally once daily for up to 34 weeks. Participants received filgotinib 200 mg in the Main Study.
Arm/Group | Filgotinib 200 mg (Main Study) | Filgotinib 100 mg (Main Study) | Adalimumab 40 mg (Main Study) | Placebo (Main Study) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) | Filgotinib 200 mg From Adalimumab 40 mg (LTE) | Filgotinib 100 mg From Adalimumab 40 mg (LTE) | Filgotinib 200 mg From Placebo (LTE) | Filgotinib 100 mg From Placebo (LTE)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/9 | 0/20 | 0/4 | 0/3 | 0/1 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19 | 0/9 | 0/20 | 0/4 | 0/3 | 0/1 | 0/1 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 4/19 | 7/19 | 2/9 | 9/20 | 1/4 | 0/3 | 0/1 | 0/1 | 1/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (Main Study) (N=19) | Filgotinib 100 mg (Main Study) (N=19) | Adalimumab 40 mg (Main Study) (N=9) | Placebo (Main Study) (N=20) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) (N=4) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) (N=3) | Filgotinib 200 mg From Adalimumab 40 mg (LTE) (N=1) | Filgotinib 100 mg From Adalimumab 40 mg (LTE) (N=1) | Filgotinib 200 mg From Placebo (LTE) (N=2) | Filgotinib 100 mg From Placebo (LTE) (N=2)
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (Main Study) (N=19) | Filgotinib 100 mg (Main Study) (N=19) | Adalimumab 40 mg (Main Study) (N=9) | Placebo (Main Study) (N=20) | Filgotinib 200 mg From Filgotinib 200 mg (LTE) (N=4) | Filgotinib 100 mg From Filgotinib 100 mg (LTE) (N=3) | Filgotinib 200 mg From Adalimumab 40 mg (LTE) (N=1) | Filgotinib 100 mg From Adalimumab 40 mg (LTE) (N=1) | Filgotinib 200 mg From Placebo (LTE) (N=2) | Filgotinib 100 mg From Placebo (LTE) (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of the study and insufficient number of participants enrolled, all the hypothesis testing performed and the p values reported were nominal. Therefore, the results need to be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04115748/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04115748/SAP_001.pdf